CLINICAL TRIAL: NCT07097090
Title: Inclusion 4 Children (Https://inclusion4children.it)
Brief Title: Improving Emotion Recognition Ability to Support Social Development in Children: A Quasi-Experimental Study
Acronym: I4C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Alessandro De Santis, Inclusion 4 Children, University of Foggia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 43681
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2023-01

CONDITIONS: Emotions; Facial Emotion Recognition; Antisocial Behavior; Nonverbal Communication; Intelligence
Keywords: Emotion Recognition Ability; Prosocial Behavior; Nonverbal Intelligence; Primary School Children
MeSH Terms: conditions — Antisocial Personality Disorder; Nonverbal Communication; Altruism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion Recognition Training Group (Experimental)
  Interventions: Behavioral: Emotion Recognition Training Program: A structured school-based intervention designed to enhance children's ability to recognize emotions through facial expressions, tone of voice, and body language.
- No Intervention Control Group (Active Comparator)
  Interventions: Behavioral: No Intervention: Observational Cohort

INTERVENTIONS:
Behavioral: Emotion Recognition Training Program: A structured school-based intervention designed to enhance children's ability to recognize emotions through facial expressions, tone of voice, and body language. — Emotion Recognition Training Program Integrated CASEL-based activities with CBT principles and digital tools to enhance emotional attribution and recognition in primary school children.
  The intervention consisted of three structured activities based on the CASEL framework (Collaborative for Academic, Social, and Emotional Learning), integrated with cognitive-behavioral principles inspired by the model of Albert Ellis. Sessions included interactive use of digital whiteboards and narrative tools (e.g., emotion-themed interactive stories), aimed at improving children's ability to attribute emotions to others and to emotionally evaluate events.
  In addition, a neurostimulative component was included, exposing children to visual stimuli with either neutral or fear-inducing emotional valence. Participants were asked to rate the perceived emotional intensity, supporting the development of self-regulation and emotional differentiation.
  Arms: Emotion Recognition Training Group
Behavioral: No Intervention: Observational Cohort — Control group received no intervention in order to serve as a baseline for comparison, isolating the effects of the emotion recognition training on behavioral and cognitive outcomes.
  Arms: No Intervention Control Group

SUMMARY:
The goal of this quasi-experimental study is to investigate whether enhancing emotion recognition abilities can improve social behavior in primary school children. The study focused on children aged approximately 6 to 9 years (both sexes), attending elementary school, without neurological or psychiatric diagnoses.

The main questions it aims to answer are:

Is there an inverse relationship between children's ability to recognize nonverbal emotional cues and antisocial behavior, as assessed by teachers?

Does nonverbal intelligence (measured through Raven's Colored Progressive Matrices) significantly predict emotion recognition ability (ERA)?

Researchers compared a group of children who received the intervention (experimental group) with a control group that did not, to see whether improvements in ERA relate to higher prosocial behavior and fewer behavioral difficulties.

Participants were asked to:

Complete the DANVA-2-RV, a standardized tool to assess nonverbal emotion recognition, updated and validated on the study sample;

Complete Raven's Colored Progressive Matrices, to measure nonverbal IQ;

Have their behavior assessed via the SDQ - Teacher Version, filled out by their classroom teachers.

A total of 140 children from four schools were enrolled. Participants were assigned non-randomly to an experimental or control group. Six teachers were involved in the behavioral assessments.

The study is concluded. Expected outcomes include:

A negative correlation between prosocial behavior and emotional confusion;

A weak or non-significant relationship between nonverbal intelligence and emotion recognition ability.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in primary school (ages 6-9)
* Parental/guardian informed consent obtained
* Teacher agreement to complete SDQ - Teacher Version
* Availability for participation in both pre- and post-assessment sessions
* No diagnosed cognitive, psychiatric, or neurological disorders

Exclusion Criteria:

* Documented diagnosis of neurodevelopmental disorders (e.g., ASD, ADHD, intellectual disability)
* Severe visual, auditory, or motor impairments affecting test participation
* Incomplete parental consent or teacher refusal to collaborate
* Absence from school during key phases of assessment

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Emotion Recognition Accuracy Between Groups | Pre-test at Month 0, Intervention begins at Month 6, Post-test at 3 months after intervention (Month 9)
  Measured using the DANVA-2-RV. Emotion recognition accuracy scores (correct identification of basic emotions) will be compared between the intervention and control groups.

SECONDARY OUTCOMES:
Cross-Sectional Observation of Behavioral Profiles | Single time point at study entry (Month 0).
  Observation of behavioral difficulties and prosocial behaviors (via SDQ - Teacher Version).
Cross-Sectional Observation of Cognitive Profiles | Single time point at study entry (Month 0).
  Observation of nonverbal intelligence (via Raven's Colored Progressive Matrices).

CONTACTS AND LOCATIONS:
Locations (1):
- Alessandro De Santis, Foggia, Apulia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Due to the involvement of children in a protected age range, the dataset contains sensitive information that cannot be publicly shared in its raw form. However, the research team is willing to provide de-identified and anonymized data upon reasonable request, ensuring that all personally identifiable or sensitive details are masked in accordance with ethical standards and institutional policies.

REFERENCES:
- [Background] Naumann S, Bayer M, Kirst S, van der Meer E, Dziobek I. A randomized controlled trial on the digital socio-emotional competence training Zirkus Empathico for preschoolers. NPJ Sci Learn. 2023 Jun 19;8(1):20. doi: 10.1038/s41539-023-00169-8. PMID 37336872
- [Background] Wells AE, Hunnikin LM, Ash DP, van Goozen SHM. Children with Behavioural Problems Misinterpret the Emotions and Intentions of Others. J Abnorm Child Psychol. 2020 Feb;48(2):213-221. doi: 10.1007/s10802-019-00594-7. PMID 31686284
- [Background] Collaborative for Academic, Social, and Emotional Learning (CASEL). CASEL Guide to Schoolwide SEL Implementation. Chicago, IL: CASEL; 2020.
- [Background] Song JH, Colasante T, Malti T. Helping yourself helps others: Linking children's emotion regulation to prosocial behavior through sympathy and trust. Emotion. 2018 Jun;18(4):518-527. doi: 10.1037/emo0000332. Epub 2017 Jun 5. PMID 28581324
- [Background] Izard C, Fine S, Schultz D, Mostow A, Ackerman B, Youngstrom E. Emotion knowledge as a predictor of social behavior and academic competence in children at risk. Psychol Sci. 2001 Jan;12(1):18-23. doi: 10.1111/1467-9280.00304. PMID 11294223
- See also: Related Info — https://inclusion4children.it